CLINICAL TRIAL: NCT04349605
Title: Meditation and Yoga for Patients With Persistent Symptoms After Lyme Disease
Brief Title: Meditation and Kundalini Yoga for Persistent Lyme-related Symptoms - an Online Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn given new information indicating a new study design would be preferable
Sponsor: Research Foundation for Mental Hygiene, Inc. (Other)
Responsible Party: Principal Investigator, Brian A Fallon, Professor of Psychiatry, Research Foundation for Mental Hygiene, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7613
Record Dates: First submitted 2020-04-14; First posted 2020-04-16 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Post-Treatment Lyme Disease
Keywords: Lyme disease; Kundalini Yoga; Meditation; Chronic Lyme Disease
MeSH Terms: conditions — Post-Lyme Disease Syndrome; Lyme Disease | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of the three treatment arms of the study - Kundalini Yoga, Meditation, or Treatment as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Meditation (Experimental): This is a daily 15 minute meditation with guided breathing. Accessible through an app.
  Interventions: Behavioral: Meditation
- Kundalini Yoga (Experimental): This is a daily 30 minute practice of Kundalini Yoga (stretching, guided breathing, and meditation). Accessible by smart phone, tablet or computer.
  Interventions: Behavioral: Kundalini Yoga
- Treatment as Usual (No Intervention): This group will serve as the comparison to assess the efficacy of the active treatments in that no study treatment will be provided. The participants will be asked to not start new treatments during the 8 weeks of the study.

INTERVENTIONS:
Behavioral: Meditation — Meditation involves guided breathing and mindfulness training.
  Arms: Meditation
Behavioral: Kundalini Yoga — Kundalini Yoga involves stretching, guided breathing and meditation
  Arms: Kundalini Yoga

SUMMARY:
This randomized, controlled study examines whether a daily practice over 8 weeks of Kundalini Yoga or Meditation can help to reduce pain and/or fatigue among patients with symptoms that persist despite prior antibiotic treatment.

DETAILED DESCRIPTION:
Research reports indicate that approximately 5-20% of patients treated for Lyme disease with the IDSA-recommended 2-4 week course of antibiotics will continue to have symptoms of fatigue, pain, cognitive problems, and/or joint and muscle aches despite prior antibiotic treatment. The symptoms can last months to years after treatment. The medical community officially calls this condition "Post-treatment Lyme disease Syndrome" (PTLDS) when patients meet strict inclusion and exclusion criteria. The patient community commonly calls this condition "chronic Lyme disease" (CLD). Although there is debate about the exact cause of these symptoms, there is widespread agreement that this is a growing public health problem as an increasing number of patients are suffering with symptoms of pain, fatigue, and cognitive problems ("brain fog") despite having received not just the standard treatment courses but even after many courses of antibiotics and other interventions.

While antibiotic therapy is the key to the treatment of active infection, other approaches are needed for those patients whose symptoms persist despite the best antibiotic treatment efforts. Alternative treatments that can assuage fatigue, muscle and joint pains, and improve cognitive function are urgently needed. Recent studies indicate that mind body practices (e.g., meditation; Kundalini Yoga) can be helpful strategy in reducing chronic symptoms, such as pain, fatigue, and poor mental focus. This study examines the efficacy of two mind-body therapies among patients with PTLDS and CLD: a) the breathing, meditation, and stretching techniques common to Kundalini Yoga practice; and b) meditation and breathing techniques common to Western meditation practices. We plan to assess the degree to which these practices can reduce the chronic symptoms compared to a wait-list control group. Because fatigue and multi-system symptoms are so common among patients with PTLDS or CLD, these will be the primary focus of this study. Primary outcome will be improvement in these self-reported core symptoms and in self-reported quality of life. Secondary outcomes will assess cognitive complaints, pain, physical and mental functioning, somatic symptoms, and psychopathology.

This will be an on-line study. During this study, patients will be screened through an on-line process, review consent, and complete self-report questionnaires. 225 patients will be enrolled. Of these, 75 will be randomly assigned to Kundalini yoga and meditation therapy, 75 will be assigned to a meditation & mindfulness App, and 75 will be assigned to a "treatment as usual" wait-list. Assessments will be conducted weekly for 8 weeks; there will also be a 6 month follow-up by questionnaire. Study participants randomized to the "treatment as usual" control group will be offered the option of receiving guided on-line meditation at the end of the 8 weeks.

Should this study find evidence suggesting that either meditation therapy and/or Kundalini Yoga are helpful in reducing the symptoms that persist after Lyme disease treatment, this would be a valuable and welcome research finding.

ELIGIBILITY:
Inclusion Criteria:

1. Continued Lyme disease-related symptoms despite prior antibiotic treatment
2. Current symptoms of either fatigue or pain that is moderate in severity
3. Treatment history over the prior 8 weeks: Either no treatment or it's been stable
4. Willingness to not start a new medical or psychiatric treatment during the 8 study weeks
5. Access to a smart phone
6. Age 18-70 and able to read and understand English
7. Lives in the United States

Exclusion Criteria:

1. Current severe depression, Substance abuse in the last 6 months, pain disorder treated with an opiate-based medication, or current or past episodes of Psychosis or Bipolar disorder.
2. Individuals with physical disability that might make study participation difficult.
3. Individuals whose current medical status is so severe or unstable that participation in the study (and not receiving new treatments from other providers) would be difficult
4. Unwillingness to complete questionnaires on-line or dedicate thirty minutes daily to meditation and/or stretching
5. Unwillingness to continue in the study for 8 weeks by completing self-report evaluations if randomly assigned to the wait-list rather than to Kundalini Yoga or Meditation.
6. Individuals unwilling to delay starting any new Mind-body practice (e.g., meditation , Yoga) until after the 8 weeks of the study have been completed.
7. Individuals with a current daily practice of Mindfulness-based stress reduction or those who currently have a daily practice of meditation or yoga
8. Individuals unwilling to provide records of prior diagnosis and treatment for Lyme disease
9. Individuals unwilling to accept push notifications to their smartphone or computer

   -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-20 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | Up to 24 weeks
  A Fatigue impact measure
General Symptom Questionnaire-30 | Up to 24 weeks
  A self-report measure of multi-system symptom burden
Quality of Life Experience Scale | Up to 24 weeks
  A measure of qualify of life

SECONDARY OUTCOMES:
Pain Visual Analog Scale | Up to 24 weeks
  A self-report measure of pain severity
Applied Cognition scale | Up to 24 weeks
  A self-report measure of cognitive function
PROMIS-29 | Up to 24 weeks
  A self-report measure of seven symptom and functional domains
SF-12 | Up to 24 weeks
  A self-report measure of physical and mental functioning

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Fallon, MD, Principal Investigator — Columbia University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carlson LE, Garland SN. Impact of mindfulness-based stress reduction (MBSR) on sleep, mood, stress and fatigue symptoms in cancer outpatients. Int J Behav Med. 2005;12(4):278-85. doi: 10.1207/s15327558ijbm1204_9. PMID 16262547
- [Background] Grossman P, Kappos L, Gensicke H, D'Souza M, Mohr DC, Penner IK, Steiner C. MS quality of life, depression, and fatigue improve after mindfulness training: a randomized trial. Neurology. 2010 Sep 28;75(13):1141-9. doi: 10.1212/WNL.0b013e3181f4d80d. PMID 20876468
- [Background] Khalsa MK, Greiner-Ferris JM, Hofmann SG, Khalsa SB. Yoga-enhanced cognitive behavioural therapy (Y-CBT) for anxiety management: a pilot study. Clin Psychol Psychother. 2015 Jul-Aug;22(4):364-71. doi: 10.1002/cpp.1902. Epub 2014 May 7. PMID 24804619
- [Background] Shannahoff-Khalsa D, Fernandes RY, Pereira CAB, March JS, Leckman JF, Golshan S, Vieira MSR, Polanczyk GV, Miguel EC, Shavitt RG. Kundalini Yoga Meditation Versus the Relaxation Response Meditation for Treating Adults With Obsessive-Compulsive Disorder: A Randomized Clinical Trial. Front Psychiatry. 2019 Nov 11;10:793. doi: 10.3389/fpsyt.2019.00793. eCollection 2019. PMID 31780963
- [Background] Wang YY, Li XH, Zheng W, Xu ZY, Ng CH, Ungvari GS, Yuan Z, Xiang YT. Mindfulness-based interventions for major depressive disorder: A comprehensive meta-analysis of randomized controlled trials. J Affect Disord. 2018 Mar 15;229:429-436. doi: 10.1016/j.jad.2017.12.093. Epub 2018 Jan 3. PMID 29331704